CLINICAL TRIAL: NCT06219239
Title: Evaluation of the Safety and Efficacy of KL003 Gene Therapy in Patients With Transfusion-dependent β-thalassemia With No Conditioning Regimen
Brief Title: Safety and Efficacy of the Lentiviral Vector in Gene Therapy of Beta-thalassemia Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Collaborators: Kanglin Biotech (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2023084
Record Dates: First submitted 2024-01-05; First posted 2024-01-23 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-03

CONDITIONS: Transfusion-dependent Beta-Thalassemia
Keywords: Beta-Thalassemia; Hematopoietic Stem-Cell Transplantation; KL003; Gene therapy; no conditioning regimen
MeSH Terms: conditions — beta-Thalassemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- KL003 cell injection Drug Product (Experimental): Traditional myeloablative conditioning regimen consists of Busulfan, which may increase the risk of irreversible pulmonary fibrosis, VOD, and infertility due to potential serious toxicity. In this study, we intend to use genetic hematopoietic stem cells (lentivirus transduction) transfusion with no conditioning regimen, which could avoid toxicity due to chemotherapy drugs.
  Interventions: Genetic: KL003 cell injection Drug Product

INTERVENTIONS:
Genetic: KL003 cell injection Drug Product — No conditioning regimen for transfusion of auto-HSC transduced with lentiviral vector encoding βA-T87Q-globin gene

SUMMARY:
This is a non-randomized, open-label, single-dose study. The aim of this study is to evaluate the safety and efficacy of the treatment with lentiviral vector encoding βA-T87Q-globin gene transduced autologous hematopoietic stem cells transfusion in subjects with transfusion-dependent β-thalassemia.

ELIGIBILITY:
Inclusion Criteria:

* Male or female age between 3-35 years
* Diagnosis of transfusion-dependent β-thalassemia and a history of at least 100 mL/kg/year of pRBCs or ≥8 transfusions of pRBCs per year for the prior 2 years
* Documented baseline, or pretransfusion, Hb level≤7 g/dL
* Karnofsky performance status ≥70 for subjects≥16 years of age; Lansky performance status of ≥70 for subjects<16 years of age
* Eligible to undergo auto-HSCT
* Willing and able to follow the research procedures and conditions, with good compliance
* Willing to receive at least the 2 years follow-up and maintain detailed medical records, including transfusion history
* Subject and/or legal guardians voluntarily participated in this clinical trial and signed the informed consent form, and can complete all follow-ups in accordance with the protocol requirements

Exclusion Criteria:

* Presence of clear contraindications for hematopoietic stem cell collection
* Diagnosis of composite α thalassemia
* A white blood cell (WBC) count <3×10^9/L, and/or platelet count <100×10^9/L not related to hypersplenism
* Subjects with severe iron overload at the time of screening: severe iron overload of the liver showed by MRI, serum ferritin ≥ 5000 ng/mL, or moderate to severe iron overload of the heart
* Any prior or current malignancy or myeloproliferative or significant immunodeficiency disorder
* Meet the criteria for allo-HSCT and with an identified willing donor with a full HLA match
* Prior receipt of gene therapy or allo-HSCT
* Subjects with any severe active fungal, bacterial, viral, tuberculosis or other infection, including active hepatitis B (defined as serum HBV-DNA ≥2000 IU/ml), active hepatitis C virus, HCV) infection, human immunodeficiency virus (HIV) antibody-positive or active syphilis patients, etc.
* Immediate family member (i.e. parent or siblings) with a known Familial Cancer Syndrome (including but not limited to hereditary breast and ovarian cancer syndrome, hereditary non-polyposis colorectal cancer syndrome and familial adenomatous polyposis)
* Diagnosis of a significant psychiatric disorder of the subject that could seriously impede the ability to participate in the study
* History of major organ damage including:

  1. Liver function test suggest AST or ALT levels >3× upper limit of normal (ULN);
  2. Total serum bilirubin value >2.5×ULN;if combined with Gilbert syndrome, total bilirubin >3×ULN and direct bilirubin value >2.5×ULN;
  3. History of bridging fibrosis, cirrhosis;
  4. Left ventricular ejection fraction <45%;
  5. New York Heart Association (NYHA) class III or IV congestive heart failure;
  6. Severe arrhythmia requiring medical treatment;
  7. Uncontrolled hypertension or unstable angina pectoris;
  8. Myocardial infarction or bypass or stent surgery within 12 months before drug administration;
  9. Valvular disease with clinical significance;
  10. Baseline calculated eGFR<60mL/min/1.73m2;
  11. Pulmonary function: FEV1/FVC<60% and/or diffusion capacity of carbon monoxide (DLco) <60% of prediction;
  12. Evidence of clinically significant pulmonary hypertension requiring medical intervention.
* Uncorrectable coagulation dysfunction or history of severe bleeding disorder
* Any other condition that would render the subject ineligible for HSCT, as determined by the attending transplant physician
* Known allergy to clinical trial drug (plerixafor or G-CSF or busulfan) or ingredient(DMSO etc.)
* Participated in other clinical studies within 3 months prior to screening
* Inoculated live vaccine within 6 weeks prior to screening
* Pregnancy or breastfeeding women; Subjects or their sexual partners were unable to take medically recognized effective contraceptive measures during the 27-month study period
* The subjects or their parents would not comply with the study procedures outlined in the protocol
* The subjects received hydroxyurea or thalidomide or hypomethylating drugs within 3 months before hematopoietic stem cell collection
* Patients considered to be ineligible for the study by the investigator for reasons other than the above

Ages: 3 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 3 (Estimated)
Dates: Start 2024-01-04 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The number, frequency and severity of adverse events (AE) after reinfusion of KL003 drug products | within 6 months
The proportion of participants who meet the definition of transfusion independence (TI) for at least 6 months | Up to 24 months post transplant
  TI is defined as Hb ≥ 90.0 g/L after reinfusion and without disease-related routine blood transfusion for 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Hematology & Blood Diseases Hospital, Tianjin, Tianjin Municipality, China